CLINICAL TRIAL: NCT06370390
Title: Community-based Group Rehabilitation Program for Stroke Patients With Dysphagia: a Randomized Controlled Trial
Brief Title: Community-based Group Rehabilitation Program for Stroke Patients With Dysphagia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copka Sonpashan (Other Government)
Responsible Party: Sponsor-Investigator, Copka Sonpashan, Research Director, Chao Phya Abhaibhubejhr Hospital
Organization: Chao Phya Abhaibhubejhr Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: community - stroke dysphagia
Record Dates: First submitted 2024-04-13; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Experimental): Patients in the intervention group received swallowing function training in community public spaces for 5 days every week for a 4-week period.
  Interventions: Behavioral: swallowing function training
- The control group (No Intervention): No intervention will be applied

INTERVENTIONS:
Behavioral: swallowing function training — The group rehabilitation program comprised daily 60-minute sessions, five times per week for a duration of 4 weeks.
  The group rehabilitation program included: Rehabilitation oral and facial exercises, Game-based surface electromyographic biofeedback training, Participants experience sharing, Individual direct feeding training
  Arms: the intervention group

SUMMARY:
Community-based exercise programs have demonstrated potential for implementation in older adults; however, it remains imperative to ascertain whether this strategy will yield comparable benefit in stroke patients with dysphagia.Participants were randomly assigned to either the intervention group or the control group. Patients in the intervention group received swallowing function training in community public spaces for 5 days every week for four-week period (60 minutes per day). Patients in the control group received no intervention. Penetration-Aspiration Scale and Standardized Swallowing Assessment (SSA), depressive symptoms (Geriatric Depression Scale-15), and meal duration were assessed before and after all the treatment.

DETAILED DESCRIPTION:
Stroke is complicated by oropharyngeal dysphagia in 29 to 81% of patients. Up to 40% of these individuals continue to experience swallowing difficulty even after a year later, which is associated with an increased risk of consequences such as aspiration pneumonia, dehydration, and malnutrition.

Community-based exercise programs have demonstrated potential for implementation in older adults; however, it remains imperative to ascertain whether this strategy will yield comparable benefit in stroke patients with dysphagia.Participants were randomly assigned to either the intervention group or the control group. Patients in the intervention group received swallowing function training in community public spaces for 5 days every week for four-week period (60 minutes per day). Patients in the control group received no intervention. Penetration-Aspiration Scale and Standardized Swallowing Assessment (SSA), depressive symptoms (Geriatric Depression Scale-15), and meal duration were assessed before and after all the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age over 65 years old.
* No hospitalization within the past six months.
* With clear consciousness and able to cooperate with questionnaires and training.
* The elderly people who voluntarily participate and agree to adhere until the end of the study.
* early dysphagia.

Exclusion Criteria:

* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Physical disability.
* Simultaneously receiving other therapies that might influence this study.
* Individuals with a gastrostomy.
* Abnormalities of the oral, pharyngeal, or esophageal structures.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Standardized Swallowing Assessment Scale | day 1 and day 28
  The Standardized Swallowing Assessment Scale is a commonly used tool for evaluating swallowing function. It is widely applied in medical and rehabilitation fields to assess an individual's swallowing ability and the smooth passage of food/liquid through the esophagus. The scale ranges from 18 to 46, with lower scores indicating better swallowing function.

SECONDARY OUTCOMES:
Time consumed in eating | day 1 and day 28
  The investigators require participants to eat a lunch according to their daily intake and habits, and count the time consumed
Penetration-Aspiration Scale | day 1 and day 28
  Penetration-Aspiration Scale was used to assess dysphagia under Videofluoroscopic Swallowing Study, primarily evaluating the extent to which fluid food entered the airway and caused penetration or aspiration during the swallowing process. As the level increased, the severity of dysphagia also increased.
15-item Geriatric Depression Scale | day 1 and day 28
  The 15-item Geriatric Depression Scale (GDS-15) is a widely used screening tool designed to detect depression in elderly individuals aged 65 and older.Scores on the GDS-15 range from 0 to 15, with higher scores indicating a higher likelihood of depression. A cutoff score of 5 or higher is commonly used to indicate possible depression, although this may vary depending on the population being assessed and the purpose of the screening.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Wi, Principal Investigator — Site Coordinator of United Medical Group located in Miami